CLINICAL TRIAL: NCT05255744
Title: Assessment of the Seal, Comfort, Usability and Performance of the Prototype Whitsundays Nasal Mask System in the Singapore Home Environment
Brief Title: Whitsundays (Nasal) Singapore External Clinical Study 1 Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ResMed (Industry)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SLP-21-11-01
Record Dates: First submitted 2021-12-14; First posted 2022-02-24 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a randomized, open label, cross over study to evaluate the Whitsundays nasal mask system (prototype mask) against a released mask system, the ResMed AirFit N30i Quiet mask system.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Whitsundays nasal mask (Experimental): Participants will be asked to take home the investigational mask to use at night while they sleep in place of their own mask. The participant's therapy and comfort settings will not be altered.
  Interventions: Device: Positive Airway Pressure (PAP) Therapy
- AirFit N30i Quiet mask (Active Comparator): Participants will be asked to take home the comparator mask to use at night while they sleep in place of their own mask. The participant's therapy and comfort settings will not be altered.
  Interventions: Device: Positive Airway Pressure (PAP) Therapy

INTERVENTIONS:
Device: Positive Airway Pressure (PAP) Therapy — PAP therapy supplies pressurized air from the flow generator to the upper airway via air tubing and a mask to prevent the repetitive collapse of the upper airway during sleep.

SUMMARY:
Each Whitsunday mask or AirFit N30i Quiet mask is worn for 7 nights. The overall purpose of this study is to evaluate the performance of the Whitsundays nasal mask system (a prototype mask) compared to the ResMed AirFit N30i Quiet mask system (a benchmark mask) in relation to seal, comfort, usability, overall performance, and efficacy.

DETAILED DESCRIPTION:
This is a randomized, open label, cross over study to evaluate the Whitsundays nasal mask system (prototype mask) against a released mask system, the ResMed AirFit N30i Quiet mask system.

The Whitsundays nasal mask system will be compared with a released mask, ResMed's AirFit N30i Quiet, as it is also a nasal mask and the most appropriate benchmark. Study participants are experienced with CPAP masks and devices and therefore will use their experience to identify areas for potential improvement.

Recruitment will be done via phone calls/ SMS messages/ emails <TBC with PI>. Participants will be explained the details of the trial and those who wish to take part will be invited to a selected site for the first study visit.

Visit 1: Participants will provide written informed consent. Participants will be shown the mask systems and trial them for fit and comfort. Participants may be asked initial questions on their first thoughts on the mask systems. If the participant and assessor are happy to proceed, the participants will use the mask and loan CPAP for trial.

Visit 2: After trialing the mask systems, participants will be asked to complete a questionnaire regarding the seal and comfort of the mask system(s). Participants will then take the second mask system home to test.

Visit 3: The participant will return the masks and CPAP device to the assessor. The participants' questionnaire responses will be reviewed. This concludes the participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients willing to give written informed consent
* Patients who can read and comprehend English
* Patients who ≥ 21 years of age
* Patients being treated for OSA with PAP therapy for ≥ 6 months
* Patients currently using a suitable mask system (any nasal mask )
* Patients who can trial the masks for up to 7 nights each

Exclusion Criteria:

* Patients using Bilevel flow generators
* Patients who are or may be pregnant
* Patients with a preexisting lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury.
* Patients believed to be unsuitable for inclusion by the researcher

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-28 (Estimated); Primary Completion 2024-05-06 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Subjective usability | 6 weeks
  Comparison of the seal, comfort, usability and overall preference of the Whitsundays nasal mask system to the AirFit N30i Quiet mask system and/or Criterion Score of 6
Apnea Hypopnea Index (Events/hour) | 6 weeks
  Objective AHI taken from the participant's CPAP device used during the trial, with a comparison of the Whitsundays nasal mask to the benchmark AirFit N30i Quiet mask or clinically relevant data. nasal mask system to the AirFit N30i Quiet mask system and/or Criterion Score of 6

SECONDARY OUTCOMES:
General Usability | 6 weeks
  General subjective usability scores from participant. Each usability items of the Whitsundays Nasal Mask System and AirFit N30i Quiet Mask System will be rated on a Likert Scare questionnaire. A score of 10 is considered very favourable whereas score of 0 is considered very unfavourable.
Leak (L/minute) | 6 weeks
  Calculated leak from the CPAP device provides information on how well the Whitsundays Nasal Mask and AirFit N30i Quiet Mask fit on the patient.
CPAP Pressure (cmH2O) | 6 weeks
  Calculated average pressure from the CPAP device, which indicates how much pressure patients need to keep the airway open.
Usage Hours (hours/night) | 6 weeks
  Average usage hours taken from the participants' CPAP device used during the study.

IPD SHARING:
Plan to Share IPD: No